CLINICAL TRIAL: NCT06443905
Title: Efficacy, Safety and Cost-effectiveness of Xueshuantong Injection (Lyophilized) in the Prevention of Venous Thromboembolism (VTE) in Hospitalized Patients at Risk of Bleeding: a Real-world Cohort Study
Brief Title: Xueshuantong Injection (Lyophilized) in the Prevention of Venous Thromboembolism (VTE) in Hospitalized Patients
Status: Active, not recruiting | Type: Observational
Sponsor: China-Japan Friendship Hospital (Other)
Collaborators: Guangxi Wuzhou Pharmaceutical (GROUP) Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Wanmu Xie, chief physician, China-Japan Friendship Hospital
Other Study IDs: JVMID-2023101
Record Dates: First submitted 2024-04-26; First posted 2024-06-05 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-05

CONDITIONS: Venous Thromboembolism (VTE); Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism; Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- PNS_ONLY: Only Xueshuantong injection(lyophilized) is used after surgery
- NON_INT: No thrombus prophylaxis after surgery
- LMWH_ONLY: Only low molecular weight heparin(LMWH) is used after surgery
- PNS+LMWH: Xueshuantong injection (lyophilized) and low molecular weight heparin are used simultaneously after surgery
- ICH_CTL: Conventional treatment
- ICH_PNS: Conventional treatment + Xueshuantong injection (lyophilized)
- AIS_CTL: Conventional treatment
- AIS_PNS: Conventional treatment + Xueshuantong injection(lyophilized)

SUMMARY:
The purpose of this study is to explore the efficacy, safety and cost-effectiveness of Xueshuantong (lyophilized) for the prevention of venous thromboembolism (VTE) in patients at risk of bleeding.

DETAILED DESCRIPTION:
This is a non-randomized, observational study.

This study primarily aims to investigate the efficacy, safety, and cost-effectiveness of using Xueshuantong injection (lyophilized) for preventing venous thromboembolism (VTE) in patients susceptible to bleeding. The subjects of the study comprise patients during the perioperative period (undergoing procedures lasting 45 minutes or longer), patients with a confirmed spontaneous cerebral hemorrhage (ICH), and patients with a confirmed acute ischemic stroke (AIS).

Additional objectives of this study including:

1. to evaluate the possible dose-dependency of Xueshuantong injection (lyophilized);
2. to evaluate the impact in coagulation function after administration of Xueshuantong injection (lyophilized)

ELIGIBILITY:
Inclusion Criteria:

* Men or women of ≥18 year old;
* Hospitalized between Jan 1, 2016 and Aug. 1, 2023;
* Received intravenous (IV) Xueshuantong (lyophilized) for ≥3 days;
* Who also meet one of the following criteria:

  1. Perioperative patients:

     Performed any of the following surgical procedures (≥ 45 minutes in duration) during hospitalization- general surgery, orthopedic surgery, obstetrics and gynecology surgery, neurosurgery, urology surgery, cardiothoracic surgery, obesity surgery or cancer surgery;
  2. Hospitalization due to acute spontaneous cerebral hemorrhage:

     Diagnosed as cerebral hemorrhage (acute/subacute), or subarachnoid hemorrhage, with clinical manifestations such as conscious disturbance, dyskinesia, or sensory dysfunction. Presence of cerebral hemorrhage was confirmed by imaging;
  3. Hospitalization due to acute ischemic stroke:

Diagnosed as ischemic stroke, ischemic stroke (acute/subacute), cerebral infarction, or cerebral infarction (acute/subacute), acute stage or subacute stage of ischemic stroke, with clinical manifestations such as disturbance of consciousness, motor dysfunction, or sensory dysfunction. Presence of cerebral hemorrhage was confirmed by imaging.

Exclusion Criteria:

* Received any traditional Chinese medicine (TCM) that contains total saponins of panax notoginseseng (PNS) other than Xueshuantong (lyophilized);
* Females who are pregnant or breast-feeding;
* Diagnosed venous thromboembolism occurred before enrollment;
* Received intravenous thrombolytic therapy for other reasons during hospitalization;
* Received prophylactic or therapeutic doses of anticoagulants after major surgery;
* Placed vena cava filters for VTE prophylaxis before surgery;
* Received therapeutic dose of anticoagulants during the patient's hospital stay (AIS patients);

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Perioperative patients, spontaneous cerebral hemorrhage, acute ischemic cerebral infarction
Sampling Method: Non-Probability Sample
Enrollment: 21600 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of VTE | Within 14 days after admission (perioperative), within 14 days after admission (SCH), within 7 days after admission (AIS)
  Incidence of venous thromboembolism (VTE)

SECONDARY OUTCOMES:
Incidence of proximal DVT | Within 14 days after admission (perioperative), within 14 days after admission (SCH), within 7 days after admission (AIS)
  Proximal deep venous thrombosis (DVT).
Incidence of distal DVT | Within 14 days after admission (perioperative), within 14 days after admission (SCH), within 7 days after admission (AIS)
  Distal deep venous thrombosis (DVT).
Incidence of PTE | Within 14 days after admission (perioperative), within 14 days after admission (SCH), within 7 days after admission (AIS)
  Pulmonary thromboembolism (PTE).
Incidence of symptomatic VTE | Within 14 days after admission (perioperative), within 14 days after admission (SCH), within 7 days after admission (AIS)
  Symptomatic venous thromboembolism (VTE).
Incidence of non-symptomatic VTE | Within 14 days after admission (perioperative), within 14 days after admission (SCH), within 7 days after admission (AIS)
  Non-symptomatic venous thromboembolism (VTE)
Mortality | Within 14 days after admission (perioperative), within 14 days after admission (SCH), within 7 days after admission (AIS)
  Deaths of all causes.
Wound healing time | Within 14 days after admission (perioperative), within 14 days after admission (SCH), within 7 days after admission (AIS)
  Healing time after surgery
Length of stay | Within 14 days after admission (perioperative), within 14 days after admission (SCH), within 7 days after admission (AIS)
  Time from admission to discharge

CONTACTS AND LOCATIONS:
Locations (14):
- China (14):
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Dongguan Chinese Medicine Hospital, Dongguan, Guangdong
  - Foshan Hospital of Traditional Chinese Medicine, Foshan, Guangdong
  - Guangzhou Red Cross Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Liuchow, Guangxi
  - The First People's Hospital of Nanning, Nanning, Guangxi
  - The People's Hospital of Wuzhou, Wuzhou, Guangxi
  - Wuzhou Red Cross Hospital, Wuzhou, Guangxi
  - Yulin Second People's Hospital, Yulin, Guangxi
  - Hebei General Hospital, Shijiazhuang, Hebei
  - The Third Hospital of Changsha, Changsha, Hunan
  - Jingjiang Chinese Medicine Hospital, Jingjiang, Jiangsu
  - Qilu Hospital of Shandong University Dezhou Hospital, Dezhou, Shandong
  - Liaocheng People's Hospital, Liaocheng, Shandong